CLINICAL TRIAL: NCT03819062
Title: Sacral Neuromodulation as Treatment for Chronic Constipation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Jihong Chen, Assistant Professor, McMaster University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: McMasterChenC
Record Dates: First submitted 2019-01-16; First posted 2019-01-28 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: Chronic Constipation
Keywords: Constipation; spinal cord injury; back pain; High-Resolution Colonic Manometry; Anorectal Manometry
MeSH Terms: conditions — Constipation; Spinal Cord Injuries; Back Pain | interventions — Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: proof of concept
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Refractory Constipation with LLLT (Experimental): Low level laser therapy (LLLT) will be administered to patients with severe refractory chronic constipation
  Interventions: Device: Low Level Laser Therapy

INTERVENTIONS:
Device: Low Level Laser Therapy — A 3 week treatment period with 8 treatment sessions in total.
  Other Names: Sacral Neuromodulation; Photobiomodulation

SUMMARY:
The objective of this study is to study if low level laser therapy will do more good than harm for patients with severe chronic refractory constipation. It is a proof of concept study without a placebo arm.

DETAILED DESCRIPTION:
Patients will be offered the therapy if High-Resolution Colonic Manometry has shown that coordination between colon motility and recto-anal activity is abnormal and that autonomic nervous system assessment suggests a dysfunction of communication between the spinal cord autonomic nerves and the colon-rectum-anus. The therapy consists of a 3 week treatment with a total of 8 sessions of low level laser therapy. Effects will be assessed using symptom and quality of life questionnaires and physiological assessments of colon and pelvic floor function, at 4 weeks and 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients with severe chronic refractory constipation
* Must have undergone high resolution colonic manometry that shows abnormal coordination between colonic motility and ano-rectal function.

Exclusion Criteria:

* Pregnant patients
* Known malignancies in the area of treatment
* Active bleeding in area of treatment
* Active deep vein thrombosis
* When tatoos are present at area of treatment
* Patients that are light sensitive
* Patients who take NSAIDS or steroids.

Ages: 6 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-09-08 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Change in number of bowel movements/week | 12 weeks
  (significance level P<0.05 comparing before and after).

SECONDARY OUTCOMES:
Change in symptoms using the questionnaire PAC-SYM | 4 weeks
  The PAC-SYM questionnaire is a 12-item questionnaire that evaluates the severity of symptoms of constipation in 3 domains (stool, rectal, and abdominal symptoms) on a 5-point Likert scale ranging from 0 (absent) to 4 (very severe). Each domain score is the mean of the non-missing items for that domain. The total score is the mean of all non-missing items (ie, symptoms). The range of the domain or total score is 0 (response is 'absent' for each item) to 4 (response is 'very severe' for each item). A negative change from baseline indicates improvement, a positive change indicates worsening of symptoms. The minimum important difference indicating clinically significant improvement is minus 0.6 (Saito & Camilleri, 2018)
Change in symptoms using the questionnaire PAC-SYM | 12 weeks
  The PAC-SYM questionnaire is a 12-item questionnaire that evaluates the severity of symptoms of constipation in 3 domains (stool, rectal, and abdominal symptoms) on a 5-point Likert scale ranging from 0 (absent) to 4 (very severe). Each domain score is the mean of the non-missing items for that domain. The total score is the mean of all non-missing items (ie, symptoms). The range of the domain or total score is 0 (response is 'absent' for each item) to 4 (response is 'very severe' for each item). A negative change from baseline indicates improvement, a positive change indicates worsening of symptoms. The minimum important difference indicating clinically significant improvement is minus 0.6 (Saito & Camilleri, 2018)
Change in quality of life assessed by questionnaire PAC-QOL | 4 weeks
  The PAC-QOL scale is a 28-item self-report instrument designed to evaluate the burden of constipation on patients' everyday functioning and well-being. Each item is rated on a 5-point Likert scale ranging from 0 (not at all) to 4 (extremely). The instrument can be used to generate an overall score, but is also reported to assess 4 specific constipation-related domains including: 1) Worries and concerns (11 items), 2) Physical discomfort (4 items), 3) Psychosocial discomfort (8 items), and 4) Satisfaction (5 items). Each domain score is the mean of the non-missing items for that domain. The total score is the mean of all non-missing items. The range of the domain or total score is 0 (response is 'not at all' for each item) to 4 (response is 'extremely' for each item). A negative change from baseline indicates improvement, a positive change indicates worsening of symptoms. The minimum difference indicating clinically significant improvement is -0.5 (Marquis et al., 2005)
Change in quality of life assessed by questionnaire PAC-QOL | 12 weeks
  The PAC-QOL scale is a 28-item self-report instrument designed to evaluate the burden of constipation on patients' everyday functioning and well-being. Each item is rated on a 5-point Likert scale ranging from 0 (not at all) to 4 (extremely). The instrument can be used to generate an overall score, but is also reported to assess 4 specific constipation-related domains including: 1) Worries and concerns (11 items), 2) Physical discomfort (4 items), 3) Psychosocial discomfort (8 items), and 4) Satisfaction (5 items). Each domain score is the mean of the non-missing items for that domain. The total score is the mean of all non-missing items. The range of the domain or total score is 0 (response is 'not at all' for each item) to 4 (response is 'extremely' for each item). A negative change from baseline indicates improvement, a positive change indicates worsening of symptoms. The minimum difference indicating clinically significant improvement is -0.5 (Marquis et al., 2005)
Autonomic function assessment | 4 weeks
  Increase or decrease in parasympathetic reactivity in response to a change in body position from supine to standing expressed as Respiratory Sinus Arrhythmia (ln(ms2)); comparison before and after treatment
Anal spincter pressure | 4 weeks
  Anorectal manometry, measuring resting anal sphincter pressure in mmHg; comparison before and after treatment.
Change in anal sphincter pressure due to attempting defecation | 4 weeks
  Anorectal manometry, measuring change in resting anal sphincter pressure in mmHg; comparison before and after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jihong Chen, MD PhD, Principal Investigator — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Marquis P, De La Loge C, Dubois D, McDermott A, Chassany O. Development and validation of the Patient Assessment of Constipation Quality of Life questionnaire. Scand J Gastroenterol. 2005 May;40(5):540-51. doi: 10.1080/00365520510012208. PMID 16036506
- [Background] Saito YA, Camilleri M. Editorial: patient assessment of constipation-symptoms (PAC-SYM) questionnaire has a minimal important difference. Aliment Pharmacol Ther. 2018 Jan;47(1):138-139. doi: 10.1111/apt.14389. No abstract available. PMID 29226416